CLINICAL TRIAL: NCT02980783
Title: BEAM: Prospective Open Label Study to Evaluate the Effectiveness of Juvéderm® VOLIFT®™ With Lidocaine for Treatment of Dynamic Radial Cheek Line Skin Depressions
Brief Title: A Study to Evaluate the Effectiveness of Juvéderm® VOLIFT®™ With Lidocaine for Dynamic Radial Cheek Line Skin Depressions
Acronym: BEAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA-EAME-FAS-0397
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Cheek Line Depressions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Juvéderm® VOLIFT®™ with Lidocaine (Experimental): Juvéderm® VOLIFT®™ (hyaluronic acid) with Lidocaine was injected into the dynamic radial cheek line skin depressions on Day 1; volume of injection was determined by the investigator. If applicable, a touch-up of Juvéderm® VOLIFT®™ with Lidocaine was injected on Day 14.
  Interventions: Device: Juvéderm® VOLIFT®™ with Lidocaine

INTERVENTIONS:
Device: Juvéderm® VOLIFT®™ with Lidocaine — Juvéderm® VOLIFT®™ (hyaluronic acid) with Lidocaine is injected into the dynamic radial cheek line skin depressions on Day 1; volume of injection will not exceed 2 mL per side. If applicable, a touch-up of Juvéderm® VOLIFT®™ with Lidocaine will be injected on Day 14; volume will not exceed 1 mL per side.

SUMMARY:
This study will evaluate the effectiveness of Juvéderm® VOLIFT®™ with Lidocaine for dynamic radial cheek line skin depressions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of dynamic radial cheek lines
* Agrees not to make any changes to skin care routines, or to have any facial procedures or treatments during the study

Exclusion Criteria:

* Previous facial surgery, tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent dermal fillers or be planning to undergo any of these procedures during the study
* Undergone temporary facial dermal filler injections with any substance in the face in the 12 months prior to study entry
* Received botulinum toxin therapy of any serotype in any facial area within the previous 6 months agrees not to receive it during the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Kerson, Study Director — Allergan
Locations (1):
- Laboratoire DERMSCAN, Lyon, France

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Juvéderm® VOLIFT®™ With Lidocaine: Juvéderm® VOLIFT®™ (hyaluronic acid) with Lidocaine was injected into the dynamic radial cheek line skin depressions on Day 1; volume was determined by the investigator. If applicable, a touch-up of Juvéderm® VOLIFT®™ with Lidocaine was injected on Day 14.
Period: Overall Study
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Started | 53
Completed | 52
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who were treated with test product at least once.
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Improvement Rating (Improved and Not Improved) of Their Dynamic Radial Cheek Lines as Assessed by the Participant Using the Global Aesthetic Improvement Scale (GAIS)
Description: Participants graded the improvement of their dynamic radial cheek lines using the GAIS 5-point scale where -2=much worse to +2=much improved. Participants who rated their improvement as -2, -1, or 0 (much worse, worse, or no change, respectively) were grouped as Not Improved and those who rated their improvement as +1 or +2 (improved or much improved, respectively) were grouped as Improved. The percentages of participants who rated their cheek lines as Improved and Not Improved are reported.
Time Frame: Baseline (Day 1) to Day 45
Population: Per Protocol Population included all participants with no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 52
percentage of participants
  Improved | 98.1
  Not Improved | 1.9

2. Secondary Outcome: Change From Baseline in Mean Roughness (Ra) of the Radial Cheek Lines at Maximum Smile as Assessed by DERMATOP®
Description: The DERMATOP® is a fringe projection system used to measure wrinkles. The system collects 2-dimensional (2D) and 3-dimensional (3D) images and then calculates the roughness, texture, and amplitude of wrinkles. To ensure that repeat measurements are made in the same area, the angles of the camera were recorded, and a red positioning laser was used to mark the edge of the chin. In addition, a 2D picture of the baseline measurements was taken by the machine to position subsequent measurements. Measurements are presented in micrometers (μm). A negative change from Baseline (pre-treatment) indicates that the roughness of wrinkles decreased.
Time Frame: Baseline (Day 1) to Day 45
Population: Safety Population included all participants who used the test product at least one time. Number analyzed is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 53
μm
  Baseline (Day 1) | 96.6 (53.6)
  Change from Baseline at Day 45: number analyzed (Participants) | 52
  Change from Baseline at Day 45 | -24.8 (31.9)

3. Secondary Outcome: Change From Baseline in Mean Texture (Rz) of the Radial Cheek Lines at Maximum Smile as Assessed by DERMATOP®
Description: The DERMATOP® is a fringe projection system used to measure wrinkles. The system collects 2-dimensional (2D) and 3-dimensional (3D) images and then calculates the roughness, texture, and amplitude of wrinkles. To ensure that repeat measurements are made in the same area, the angles of the camera were recorded, and a red positioning laser was used to mark the edge of the chin. In addition, a 2D picture of the baseline measurements was taken by the machine to position subsequent measurements. Measurements are presented in micrometers. A negative change from Baseline (pre-treatment) indicates that the texture of wrinkles improved.
Time Frame: Baseline (Day 1) to Day 45
Population: Safety Population included all participants who used the test product at least once. Number analyzed is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 53
μm
  Baseline (Day 1) | 203.1 (72.3)
  Change from Baseline at Day 45: number analyzed (Participants) | 52
  Change from Baseline at Day 45 | -35.3 (43.6)

4. Secondary Outcome: Change From Baseline in Mean Amplitude (Rt) of the Radial Cheek Lines at Maximum Smile as Assessed by DERMATOP®
Description: The DERMATOP® is a fringe projection system used to measure wrinkles. The system collects 2-dimensional (2D) and 3-dimensional (3D) images and then calculates the roughness, texture, and amplitude of wrinkles. To ensure that repeat measurements are made in the same area, the angles of the camera were recorded, and a red positioning laser was used to mark the edge of the chin. In addition, a 2D picture of the baseline measurements was taken by the machine to position subsequent measurements. Measurements are presented in micrometers. A negative change from Baseline (pre-treatment) indicates that the amplitude of wrinkles decreased.
Time Frame: Baseline (Day 1) to Day 45
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 53
μm
  Baseline (Day 1) | 511.8 (217.8)
  Change from Baseline at Day 45: number analyzed (Participants) | 52
  Change from Baseline at Day 45 | -115.1 (129.4)

5. Secondary Outcome: Change From Baseline in Wrinkle Volume of Radial Cheek Lines at Maximum Smile
Time Frame: Baseline (Day 1) to Day 45
Population: No data was collected because wrinkle volume was not applicable.
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants by Improvement Rating (Response) of the Participants' Dynamic Radial Cheek Lines as Assessed by the Investigator Using the GAIS
Description: The investigator graded the improvement of the participant's dynamic radial cheek lines on both sides of their face using the 5-point GAIS where -2=much worse to +2=much improved. Responders are participants with a score of +1 or +2 (improved or much improved, respectively) on both sides; partial responder are participants with a score of +1 or +2 on only one side; and no-responders are participants with a score lower or equal to 0 on both sides. The percentages of responders, partial responders, and no-responders are reported.
Time Frame: Baseline (Day 1) to Day 45
Population: Per Protocol Population included all participants with no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 52
percentage of participants
  Responder | 94.2
  Partial Responder | 1.9
  No Responder | 3.8

7. Secondary Outcome: Percentage of Participants by Self-Perceived Age Category as Assessed by the Self-Perception of Age (SPA) Questionnaire
Description: The SPA questionnaire consists of one question: "How do you think your facial appearance looks compared to your age TODAY?" Participants could choose one of three possible answers: "I look my current age," "I look younger," or "I look older." The percentage of participants in the following SPA categories is reported: I look my current age, I look younger and I look older.
Time Frame: Baseline (Day 1) to Day 45
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 53
percentage of participants
  Baseline (Day) 1: I look my current age | 53
  Baseline (Day) 1: I look younger | 28
  Baseline (Day) 1: I look older | 19
  Day 45: I look my current age: number analyzed (Participants) | 52
  Day 45: I look my current age | 38
  Day 45: I look younger: number analyzed (Participants) | 52
  Day 45: I look younger | 60
  Day 45: I look older: number analyzed (Participants) | 52
  Day 45: I look older | 2

8. Secondary Outcome: Mean Score for the Level of Naturalness of the Appearance of Participants' Dynamic Radial Cheek Lines as Assessed by a Participant Questionnaire
Description: Participants were asked to indicate their level agreement with the following statement: "The treatment of my smile lines gave me a natural look." Responses were scored from 0 to 10, where 0=not at all to 10=very much.
Time Frame: Day 45
Population: Per Protocol Population included all participants with no major protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Number analyzed (Participants) | 52
units on a scale | 7.2 (2.2)

ADVERSE EVENTS:
Time Frame: Up to 59 Days after the First Injection
Arm/Group | Juvéderm® VOLIFT®™ With Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 31/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Juvéderm® VOLIFT®™ With Lidocaine (N=53)
Injection site bruising (General disorders) | 13
Injection site haematoma (General disorders) | 16
Injection site mass (General disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.